CLINICAL TRIAL: NCT03283683
Title: A Feasibility Study of the Use of Actigraphy to Determine Prognosis in Patients With Advanced Cancer
Acronym: AIPACa
Status: Completed | Type: Observational
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Shuchita Dhwiren Patel, Dr Shuchita Dhwiren Patel, Royal Surrey County Hospital NHS Foundation Trust
Other Study IDs: 16ONCN0004
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Cancer; Sleep
Keywords: rest-activity rhythm; survival; actigraphy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — On first visit (Day 1 of the study), the researcher will collect total 7.5mls (1½ teaspoons) of blood from a vein in the participant's arm. 5 mL of the venous blood sample will be sent for analysis at the Royal Surrey County Hospital of haematological and biochemical parameters, i.e. white blood cell count (WBC), neutrophil count, lymphocyte count, platelet count, urea, alanine aminotransferase (ALT), alkaline phosphatase (ALP), albumin, C-reactive protein (CRP). 2.5 mL of the venous blood sample will be sent for bio-banking at the Surrey Clinical Research Centre at the University of Surrey (for future transcriptome analysis i.e. RNA analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the use of actigraphy-derived measures to improve prognostication in patients with advanced cancer.

DETAILED DESCRIPTION:
An accurate assessment of prognosis (life expectancy) is important for cancer patients, their carers, and their health care professionals. In the case of patients / their carers, it allows them to plan for the future, and to make more informed decisions about further anti-cancer treatments, and about referral to supportive and palliative care services. However, previous research suggests that health care professionals are not particularly good at estimating prognosis, and frequently over-estimate prognosis.

The aim of this project is to assess the usefulness of measuring physical activity, and differences between daytime and nighttime physical activity, in determining prognosis in patients with cancer. Studies suggest that these measures may be useful in determining prognosis in certain groups of patients with cancer (e.g. patients receiving chemotherapy for colon / rectum cancer). However, these studies need to be repeated in patients with different types of cancer, and also patients receiving other types of treatment (including supportive and palliative care). The aim of this small scale ("feasibility") study is to determine whether or not a large scale ("definitive") study can be done.

The feasibility study will include 50 patients with cancer, who will be asked to rate their performance status (physical activity) on a well-used scale, and then to wear a watch-like device for one week that measures physical activity and sleep patterns. The researcher will collect a blood sample: some of which will be used for analysis of parameters, which have previously been identified as prognostic indicators and will collect and store some blood for future transcriptome analysis. Participants will also be asked to complete a sleep diary during the week, and a questionnaire about their symptoms at the beginning and end of the week. The study will last one week in total and is collaboration between the Royal Surrey County Hospital, and the University of Surrey (Surrey Sleep Research Centre).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients.
* Age ≥ 18 years.
* Diagnosis of locally advanced / metastatic cancer.
* No curative treatment available.
* Patient receiving supportive and palliative care.
* Negative response from palliative medicine physician to the "surprise" question (i.e. "would you be surprised if this patient were to die in the next 12 months").
* (Estimated) prognosis of > 2 weeks.

Exclusion Criteria:

* Inpatients.
* Age < 18 years.
* Diagnosis of local (non-advanced) cancer.
* Curative treatment available.
* Presence of a physical disability that affects daytime activity (e.g. metastatic spinal cord compression).
* Presence of a physical disability that affects movement of the non-dominant arm (e.g. lymphoedema).
* Cognitive impairment (clinical judgement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The number of participants in the feasibility study will be 50. Participants will be outpatients at the site, who meet all of the inclusion criteria and none of the exclusion criteria of the study (see above).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Dichotomy Index (I<O) | 7 days.
  Compares the amount of activity of the patient when in bed to when the patient is out of bed. An actigraphy-derived percentage of the activity counts, measured when the patient is in bed, that are inferior to (lower than) the median of the activity counts measured when the patient is out of bed.

SECONDARY OUTCOMES:
r24 | upto 7 days
  An actigraphy-derived 24hr correlation coefficient that reports on how reproducible the patient's activity is every 24 hours.
mean or average activity | 7 days.
  calculated as the average number of wrist movements per minute throughout the recording time

OTHER OUTCOMES:
Actigraphy-derived sleep parameters | 7 days
  Parameters during the presumed sleep phase of the circadian cycle; eg: Time in bed, sleep efficiency e.t.c
Physician ECOG-PS | Day 0 actigraphy and Day 8 actigraphy
  Physician's assessment of the patient's ECOG-Performance Status. The Eastern Cooperative Oncology Group performance scale (ECOG-PS) is a standardised measure for quantifying the functional status of patients with cancer and includes a numerical / categorical scale
Patient ECOG-PS | Day 0 actigraphy and Day 8 actigraphy
  Patient's assessment of their own ECOG-Performance Status
Memorial Symptom Assessment Scale - Short Form (MSAS-SF) | Day 0 actigraphy and Day 8 actigraphy
  The MSAS-SF is a validated symptom assessment tool that has been used extensively in oncology / palliative care research and includes questions on both physical and psychological symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Day 8 actigraphy
  This is a validated, self-rated questionnaire, which measures sleep quality and disturbances over a 1-month time period
Prognosis in Palliative Care Study predictor model (PiPS-B model) | Day 0 actigraphy
  Compare actigraphy-derived circadian / sleep parameters against other validated prognostic indicators
modified Glasgow Prognostic Score (mGPS) | Day 0 actigraphy
  Compare actigraphy-derived circadian / sleep parameters against other validated prognostic indicators

CONTACTS AND LOCATIONS:
Overall Officials: Derk-Jan Dijk, Study Director — Supervisor; Andrew Davies, Study Director — Supervisor; Shuchita D Patel, Principal Investigator — PhD student
Locations (1):
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No